CLINICAL TRIAL: NCT06937736
Title: Leistungsbewertung Durch Den Anwender. Evaluierung Des Blutglukose Monitoring Systems Contour Care Der Firma Ascensia gemäß DIN EN ISO 15197:2015
Brief Title: Performance Evaluation by the User of BGM Contour Care According to ISO 15197:2015
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut fur Diabetes Karlsburg GmbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024_002
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subject glucometer measurement (Experimental): Blood glucose measurement BGM for personal use
  Interventions: Diagnostic Test: blood glucose measurement by subject

INTERVENTIONS:
Diagnostic Test: blood glucose measurement by subject — blood glucose measurement by subject using finger tip capillary blood

SUMMARY:
Performance Evaluation by the User of the Blood Glucose Monitoring SystemContour Care in accordance with DIN EN ISO 15197:2015

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with clinical indication for blood glucose measurements (i.e. Diabetes mellitus)
* Male or female patients with hypo-, eu- or hyperglycemia
* The written informed consent had to be signed
* The volunteers must be older than 18 years
* The volunteers have legal capacity and are able to understand meaning, nature and possible consequences of the procedures involved

Exclusion Criteria:

* Pregnancy or lactation
* Acute or chronic diseases that

  * pose a risk of aggravation by the measure
  * pose a health hazard to the personnel
* A current constitution that does not allow participating in the study
* Participation in another study or activity with the blood glucose measuring system evaluated in the present study
* Application of substances listed in Appendix A of DIN EN ISO 15197:2015

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-07-23 (Actual)

PRIMARY OUTCOMES:
Analysis of system accuracy based on DIN EN ISO 15197 | Day 1
  Assessment of the analytical measurement performance of the blood glucose monitor

CONTACTS AND LOCATIONS:
Overall Officials: Eckhard Salzsieder, PhD, Study Director — Institut fur Diabetes Karlsburg GmbH
Locations (1):
- Institut für Diabetes Karlsburg GmbH, Karlsburg, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: No